CLINICAL TRIAL: NCT03454646
Title: Comparison of Therapeutic Strategies With Cholinesterase Inhibitors: Stop or Still (SOS) Trial
Brief Title: Comparison of Therapeutic Strategies With Cholinesterase Inhibitors (SOS TRIAL)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2016/27
Record Dates: First submitted 2018-02-09; First posted 2018-03-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Cholinesterase Inhibitors
MeSH Terms: conditions — Alzheimer Disease | interventions — Cholinesterase Inhibitors; Donepezil; Galantamine; Rivastigmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group randomized for continuing treatment (Experimental): Group who continues the cholinesterase inhibitors (CI). The treatment is one of the CI (donepezil, galantamine or rivastigmine) with market authorization and commercialized for more than 15 years in France. The choice of the treatment will be done by the specialist according to his habits; the specialist will monitor the treatment as usual.
  All randomised patients will then be followed-up for two years with regular assessment of judgment criteria every 6 months.
  Interventions: Drug: cholinesterase inhibitors (CI) (donepezil, galantamine or rivastigmine)
- Group randomized for stopping treatment (No Intervention): Group who stops the CI. No placebo will be given, over 2 years All randomised patients will then be followed-up for two years with regular assessment of judgment criteria every 6 months.

INTERVENTIONS:
Drug: cholinesterase inhibitors (CI) (donepezil, galantamine or rivastigmine) — The choice of the treatment will be done by the specialist according to his habits; the specialist will monitor the treatment as usual. All the recruited patients will be treated by CI according to the recommendations of the French HAS and the clinician's habits to choose the type of CI and adjust the dosage. After a 6-month period under CI treatment, patients will be classified according to the evolution of the Mini Mental State Examination (MMSE) as "non-responders" or responders.
  Responders patients will continue their treatment according to the habits of the clinician. Non-responder patients will be included in the RCT, with individual randomization in two groups: one group who stops the CI, one group who continues the CI. All randomized patients will then be followed-up for two years with regular assessment of judgment criteria every 6 months.
  Arms: Group randomized for continuing treatment

SUMMARY:
Cholinesterase inhibitors (CI) remain the only drugs with a recognized efficacy in mild to moderate Alzheimer's disease (AD) in spite of enormous research efforts. However, these drugs presented as "symptomatic treatment" of AD are considered as having only a weak effect on the course of AD. The reimbursement of these drugs is regularly challenged due to the lack of evidence for the impact of these drugs on milestones stages of AD evolution (survival without severe dementia, restriction in Basic Activities of Daily Living - BADL) and on major consequences in public health (hospitalization and institutionalization). The great majority of previous randomized controlled trials conducted with CI have had a too short duration and the end points were limited to cognition (ADAS Cog scale), IADL (Instrumental Activities of Daily Living) function and Global Impression of Change. New evidences from the DOMINO trial (1) conducted in UK, independently of the pharmaceutical industry, showed that the true effect of CI might be more to avoid or to delay the cognitive or functional decline in AD than to improve patients; the institutionalisation (2) was also delayed. However, this trial was conducted in patients with moderate to severe AD, and the interest of the drugs at the mild to moderate stage remains questionable.

The investigators have shown that a good surrogate marker of survival without severe dementia would be an increase of ADAS Cog scale of more than six points (3). A post hoc reanalysis of the pivotal RCT with two CI showed that in mild to moderate patients, CI was associated with a 15% decrease of patients with a deterioration of ADAS-Cog of more than six points in six months. Thus at the beginning of dementia the real effect of CI might be more of delaying the cognitive and functional decline, than to improve the patients. The main objective of the SOS trial is to demonstrate that the benefit of CI at the early phase of dementia is the same as at the later phase.

ELIGIBILITY:
Inclusion Criteria:

* New case of AD referring to a CMRR or MC.
* Diagnosis of probable or possible AD, defined according to the NINCDS-ARDRA criteria
* Mild to moderate stage, defined by a MMSE score above 15 at the time of pre-inclusion
* Patients with indication to CI treatment
* Patients Naïve to CI treatment
* Patients aged 50 years or more
* Menopause or effective contraception (for women)
* Affiliated person or beneficiary of a social security scheme
* Patients with AD LTI (Long Term Illeness)
* Patients agree to participate, with free, informed and written consent signed by the patient and his caregiver

Non Inclusion Criteria:

* Patients diagnosed with Lewy bodies disease, fronto-temporal dementia, or dementia from a cause other than Alzheimer Disease
* More severe stage of the disease, defined by a MMSE equal or below 15 at the time of inclusion
* Patients with contraindication to CI treatment
* Patients residing in an institution at the time of pré-inclusion or randomization
* Patients with a complete dependency for bathing and dressing at the time of pré-inclusion or randomization ( ADL de Katz, score 2/2 for the item "bathing" and/or "dressing")
* Patients under tutorship or curatorship, patients unable to express consent
* Patients with unstable severe general disease compromising the follow-up
* Patients without caregiver
* Patients included in another pharmacological trial
* Pregnant or breastfeeding women

Exclusion Criteria:

* CI responder patients for whom the MMSE score remained stable or became higher after 6 months of treatment
* Patients with complete dependency for bathing and dressing at the randomization visit
* Patients residing in an institution at the randomization visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is a combination of complete BADL dependency in bathing and dressing and/or institutionalization or death at 2 years after randomization. | at 30 months after patient's inclusion
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.

SECONDARY OUTCOMES:
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at inclusion
  Each of the components of the combined primary outcome, as defined above, analyzed separately.
  As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at 6 months
  Each of the components of the combined primary outcome, as defined above, analyzed separately.
  As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at 12 months
  Each of the components of the combined primary outcome, as defined above, analyzed separately As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at 18 months
  Each of the components of the combined primary outcome, as defined above, analyzed separately As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at 24 months
  Each of the components of the combined primary outcome, as defined above, analyzed separately As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
BADL dependency will be evaluated by the clinician using the BADL scale from Katz [17]. | at 30 months
  Each of the components of the combined primary outcome, as defined above, analyzed separately As previously demonstrated, bathing and dressing are the first ADL losses, also defined by Katz et al. as the thresholds of disability [17] [18]. A total limitation in bathing and dressing will be considered (each item is coded from 0 - no limitation, to 2 - total limitation).
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at inclusion
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at 6 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at 12 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at 18 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at 24 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Combination of complete BADL dependency in bathing and dressing and/or institutionalization or death | at 30 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
  For dependency in bathing and dressing, although it could be considered as less objective, we choose a level of total dependency, easy to assess with very low risk of misinterpretation.
Institutionalization with date of entry | at inclusion
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Institutionalization with date of entry | at 6 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Institutionalization with date of entry | at 12 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Institutionalization with date of entry | at 18 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Institutionalization with date of entry | at 24 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Institutionalization with date of entry | at 30 months
  Institutionalization with date of entry will be assessed by specialist at each follow-up time every 6 months. For patients not coming to the memory consultation, caregiver (formal and/or informal) and/or the general practitioner will be systematically contacted to obtain the information.
Death and date of death | at inclusion
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
Death and date of death | at 6 months
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
Death and date of death | at 12 months
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
Death and date of death | at 18 months
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
Death and date of death | at 24 months
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
Death and date of death | at 30 months
  Death and date of death will be assessed by contacting proxy or general practitioner. In case of lack of information the birth City Hall will be contacted to assess the vital status.
the ADL scale | at inclusion
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10 If the patient has a result of 2 at bathing and or dressing he can't be included at T0.
the ADL scale | at 6 months
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10 If the patient has a result of 2 at bathing and or dressing he can't be randomized at T6M
the ADL scale | at 12 months
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10
the ADL scale | at 18 months
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10
the ADL scale | at 24 months
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10
the ADL scale | at 30 months
  ADL DE KATZ BATHING :└-┘/2 0 bathes self completely
  1. needs help in bathing only one part of the body
  2. needs help with bathing more than one part of the body or not bathed DRESSING :└-┘ /2
  0 gets clothes and gets completely dressed without assistance
  1 gets clothes and gets dressed without assistance, except for assistance in tying shoes 2 receives assistance in getting clothes or in getting dressed, or stays partly or completely undressed TOILETING :└-┘/2 0 toileting without assistance (may use cane, walker, or wheelchair)
  1 receives assistance 2 doesn't go to room termed " toilet ". TRANSFER:└-┘/2 0 transfer without assistance (may be using cane or walker)
  1. transfer with assistance
  2. doesn't get out of bed. FEEDING :└-┘/2
  0 feeding without help
  1. need help cutting meat or buttering bread
  2. needs total help or requires parenteral feeding. TOTAL : └-┴-┘/10
the MMSE score | at inclusion
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the MMSE score | at 6 months
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the MMSE score | at 12 months
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the MMSE score | at 18 months
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the MMSE score | at 24 months
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the MMSE score | at 30 months
  The MMSE score will be assessed by the clinician, the psychologist or the speech therapist according to the habits of the center, using the French version of the MMSE (GRECO version)
the number of hospitalizations | at inclusion
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
the number of hospitalizations | at 6 months
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
the number of hospitalizations | at 12 months
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
the number of hospitalizations | at 18 months
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
the number of hospitalizations | at 24 months
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
the number of hospitalizations | at 30 months
  The number of hospitalizations will be assessed using standardized questionnaire, with date (month/year) and duration of hospitalization;
Pharmacologie treatments consumed by the patient | at inclusion
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.
Pharmacologie treatments consumed by the patient | at 6 months
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.
Pharmacologie treatments consumed by the patient | at 12 months
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.
Pharmacologie treatments consumed by the patient | at 18 months
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.
Pharmacologie treatments consumed by the patient | at 24 months
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.
Pharmacologie treatments consumed by the patient | at 30 months
  All the pharmacologie treatments consumed by the patient will be assessed, allowing to assess psychotropic drug consumption.

CONTACTS AND LOCATIONS:
Locations (31):
- France (31):
  - CHU d'Amiens Centre Mémoire Ressources Recherche, Amiens
  - CHU d'Angers Centre Mémoire Ressources Recherche, Angers
  - CHU de Bastia Centre Mémoire Ressources Recherche, Bastia
  - CHU de Besançon Centre Mémoire Ressources Recherche, Besançon
  - CHU de Bordeaux - Service de Neurologie - Centre Mémoire Ressources Recherche -, Bordeaux
  - CHRU Cavale Blanche Service de Gériatrie, Brest
  - Service de Neuropsychologie Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU Côte de Nacre Service de neurologie et CMRR, Caen
  - CHU de Clermont Ferrand Centre Mémoire Ressources Recherche, Clermont-Ferrand
  - Hôpital Pasteur Service de Neurologie, Colmar
  - CHU de Dijon- CMRR, Dijon
  - Chu de Grenoble CMRR, Neurologie, Grenoble
  - Hôpital Roger Salengro CMRR, Lille
  - CHU Limoges Service de neurologie et CMRR, Limoges
  - AP-HM, Marseille
  - CHU Montpellier Hôpital Gui de Chauliac CMRR, Montpellier
  - CHU de Nantes Clinique Neurologique Hôpital GR Laennec, Nantes
  - Institut Claude Pompidou Centre Mémoire de Ressources et de Recherche, Nice
  - APHP Hôpital Broca, Paris
  - Hôpital Universitaire de la Pitié Salpêtrière Pavillon François Lhermitte, Paris
  - APHP Groupe Hospitalier Saint Louis Lariboisière Fernand Widal CMRR, Paris
  - CHU La Milétrie Pôle de Gériatrie, Poitiers
  - CHU Reims Hôpital Maison Blanche Court Séjour Gériatrique, Reims
  - CHU de Rennes - Hôpital Pontchaillou / Service de Neurologie, Rennes
  - CHU de Rouen Hôpital Charles Nicolle Service Neurologie, Rouen
  - Chu de Saint-Etienne, CMRR, Saint-Etienne
  - Chu de Strasbourg Hôpital Ka Robertsau Pôle de Gériatrie - CMRR, Strasbourg
  - Centre de Recherche Clinique du Gérontopôle Cité de la Santé, Toulouse
  - CHRU de Bretonneau Unité de gérontopsychiatrie, Tours
  - CHU Nancy Service de Gériatrie-CMRR, Vandœuvre-lès-Nancy
  - Hospice Civil de Lyon Hôpital des Charpennes, Villeurbanne

IPD SHARING:
Plan to Share IPD: No